CLINICAL TRIAL: NCT01577316
Title: Clinical Trial to Evaluate the Immunogenicity and Safety of the 2011-2012 Vaccine Against Seasonal Influenza on Pregnant Women
Brief Title: Evaluate the Immunogenicity and Safety of the 2011-2012 Vaccine Against Seasonal Influenza on Pregnant Women
Acronym: VACINFL2011
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Laboratorios de Biologicos y Reactivos de México, S.A. de C.V. (Other)
Responsible Party: Principal Investigator, Ma. de Lourdes Garcia Garcia, Director of the Center of Research in Infectious Diseases, Instituto Nacional de Salud Publica, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CI 1059_1170
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Pregnancy; Investigation or Care in A Nonpregnant Woman
Keywords: vaccination; Influenza; Immunogenicity; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnant Woman (Experimental): Pregnant Woman
  Interventions: Biological: Seasonal influenza vaccination
- Nonpregnant women (Experimental): 2011-2012 Seasonal Influenza Vaccine (include A/California/7/2009 (H1N1)-like, A/Perth/16/2009 (H3N2)-like, and B/Brisbane/60/2008-like antigens) administered to 15ug without adjuvant, via intramuscular in pregnant and nonpregnant women.
  Interventions: Biological: Seasonal influenza vaccination

INTERVENTIONS:
Biological: Seasonal influenza vaccination — 2011-2012 Seasonal Trivalent Inactivated Influenza Vaccine (include A/California/7/2009 (H1N1)-like, A/Perth/16/2009 (H3N2)-like, and B/Brisbane/60/2008-like antigens) administered to 15ug without adjuvant, via intramuscular in pregnant and nonpregnant women.
  It is recommended that vaccines for use in the 2012-2013 influenza season (northern hemisphere winter) contain the following:
  * an A/California/7/2009 (H1N1)pdm09-like virus;
  * an A/Victoria/361/2011 (H3N2)-like virus;
  * a B/Wisconsin/1/2010-like virus.
  Other Names: Be recruited and will continue in parallel both groups

SUMMARY:
The hypothesis proposed in this study is that the 2011-2012 Seasonal Influenza Vaccine (including H3N2 and H1N1 subtypes of serotype A strain over the serotype B) administered to 15ug (without adjuvant) via intramuscular in pregnant women will be safe and immunogenic.

DETAILED DESCRIPTION:
Despite the fact that influenza vaccination of pregnant women is amply recommended, coverage of influenza vaccination is low. In general, there are few studies on safety of the vaccine to this group, particularly during the first three months of pregnancy or evaluating trivalent vaccines containing inactivated pandemic 2009 H1N1 virus. Studies are controversial regarding passage of maternal antibodies and protection to the newborn. The investigators propose to evaluate safety and immunogenicity of 2011-2012 seasonal trivalent influenza vaccine (Northern hemisphere)(containing an A/California/7/2009 (H1N1)-like virus; an A/Perth/16/2009 (H3N2)-like virus; a B/Brisbane/60/2008-like virus) produced by Sanofi Pasteur. Study design is a Phase II/III, two arm, non-randomized clinical trial. The investigators will recruit 120 pregnant women, 18 to 39 years of age, 14 to 34 week pregnant and 120 non-pregnant women. Trivalent influenza vaccine (0.5ml) will be administered IM in the deltoid zone. Participants will be observed for 30 min post-vaccination for acute adverse reactions and periodically during the 60 days post-vaccination for reactogenicity, adverse effects and severe adverse effects. Baseline and 28 day influenza antibodies will be measured by hemagglutination and microneutralization. Umbilical cord blood (10ml) will be drawn during delivery. Newborns will be followed monthly for growth and morbidity up to six months of age. If necessary, they will be referred for appropriate clinical care. Main outcome will be seroconversion and seroresponse at 28 days post vaccination. Results will be adjusted by study group and other relevant covariables.Safety will be analyzed according to type, severity and study group.

ELIGIBILITY:
I.Selection Criteria in pregnant women

I.a.Inclusion Criteria

1. Pregnant women aged 18 to 39 years
2. Have made at least one prenatal visit to confirm the pregnancy
3. Available for follow-up time
4. To be from 14 to 34 weeks of gestation
5. If recruitment is conducted between August and November 2011, patient could have
6. Received the Seasonal Influence Vaccine from previous period, but not the H1N1 vaccine
7. Agree to participate in the study and provide informed consent
8. Good health according to the clinical evaluation of the participant, confirming: heart
9. Rate less than 100', systolic blood pressure less than 140 mm Hg, and diastolic less or
10. Equal than 90 mmHg, and oral temperature less or equal than 37.4° C
11. Normal physical exam and laboratory test within 28 days prior to recruitment
12. HIV-negative test

I. b.Exclusion criteria

1. Preeclampsia or eclampsia
2. Treatment with immunosuppressive drugs
3. Receipt of blood products, 120 days prior to HIV screening
4. Receipt of immunoglobulin 60 days prior to screening for HIV
5. Have received live attenuated vaccines 30 days prior of vaccination
6. Have received inactivated vaccines within 14 days prior to vaccination
7. Treatment of latent or active tuberculosis
8. Autoimmune disease or immunodeficiency
9. Contraindication to receiving seasonal influenza vaccine
10. Vaccine side effects
11. History of angioedema.
12. Unstable asthma
13. Diabetes
14. Thyroidectomy or thyroid disease in the last 12 months
15. Idiopathic urticaria
16. Hypertension not well-controlled with treatment
17. Medically diagnosed bleeding diathesis, coagulopathy or platelet disorder
18. Active malignant tumor or in not-effective treatment
19. Asplenia
20. Allergic reaction to antibiotics
21. Guillain Barre
22. Psychiatric condition that difficult adherence to protocol

II.Selection criteria in nonpregnant woman

II. a.Inclusion criteria

* Nonpregnant woman aged 18 to 39 years
* Negative pregnancy test 24 hours prior to administration of the vaccine
* Agree to participate in the study and provide informed consent
* Good health according to the clinical evaluation of participant, confirming: heart rate
* less than 100 ', systolic blood pressure less than 140 mmHg, diastolic less than or equal
* to 90 mmHg, and oral temperature less than or equal to 37.4°C
* Normal physical exam and laboratory test within 28 days prior to recruitment
* HIV-negative test
* Agree to not get pregnant during the study and follow an effective contraceptive
* method
* Good health, determined this by history
* Receive the seasonal influenza vaccine at least two weeks prior to inclusion in this study

II. b.Exclusion criteria

* Being in treatment with immunosuppressive drugs
* Receipt of blood products, 120 days prior to HIV screening
* Receipt of immunoglobulin 60 days prior to screening for HIV
* Have received live attenuated vaccines 30 days of vaccination
* Have received inactivated vaccines within 14 days prior to vaccination
* Treatment of latent or active tuberculosis
* Autoimmune disease or immunodeficiency
* Contraindication to receiving seasonal influenza vaccine
* Vaccine side effects
* History of angioedema
* Unstable asthma
* Diabetes Type 2
* Thyroidectomy or thyroid disease requiring treatment in the past 12 months.
* Idiopathic urticaria
* Hypertension not well-controlled with treatment
* Medically diagnosed bleeding diathesis, coagulopathy or platelet disorder
* Active malignant tumor
* Convulsive condition
* Anatomic or functional asplenia
* Allergic reaction to antibiotics
* Guillain Barre
* Psychiatric condition

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | Day 28
  The results of this analysis will determine whether the vaccine provides protection based on the immunogenicity provided by the vaccine. They identify specific antibodies against influenza virus A (H1N1), will carry out the serological techniques by hemagglutination inhibition and microneutralization. The immunogenicity analysis will be measured by seroconversion and seroresponse

SECONDARY OUTCOMES:
Adverse events | 30 minutes immediate, day 1, 3, 5,7,11, 15 and 28
  Monitoring of pregnant women will be at monthly intervals until the time of the birth.
  Pregnant women and nonpregnant are going to be monitored for 30 min after vaccination to monitor immediate clinical reactions, and at 28 days after completing a self-registration of possible events associated with vaccination, as well as follow-up home visits on days 1, 3, 5, 7, 11, 15, 21, and 28.
  At day 28, will be made a complete clinical evaluation and blood sampling for assessment of immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garcia Garcia, DCs, Principal Investigator — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- National Institute of Public Health, Cuernavaca, Morelos, Mexico